CLINICAL TRIAL: NCT03761017
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation and Cohort Expansion Study of MGD019, a Bispecific DART® Protein Binding PD-1 and CTLA-4 in Patients With Unresectable or Metastatic Neoplasms
Brief Title: MGD019 DART® Protein in Unresectable/Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD019-01
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Squamous Cell Non Small Cell Lung Cancer; Prostate Cancer Metastatic; Cutaneous Melanoma; Colorectal Cancer; Advanced Cancer; Solid Tumor, Adult
MeSH Terms: conditions — Melanoma; Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Cohort 1 (Experimental): 0.03 mg/kg administered IV every 3 weeks.
  Interventions: Biological: Lorigerlimab
- Cohort 2 (Experimental): 0.1 mg/kg administered IV every 3 weeks.
  Interventions: Biological: Lorigerlimab
- Cohort 3 (Experimental): 0.3 mg/kg administered IV every 3 weeks.
  Interventions: Biological: Lorigerlimab
- Cohort 4 (Experimental): 1.0 mg/kg administered IV every 3 weeks.
  Interventions: Biological: Lorigerlimab
- Cohort 5 (Experimental): 30. mg/kg administered IV every 3 weeks.
  Interventions: Biological: Lorigerlimab
- Cohort 6 (Experimental): 6.0 mg/kg administered IV every 3 weeks.
  Interventions: Biological: Lorigerlimab
- Cohort 7 (Experimental): 10.0 mg/kg administered IV every 3 weeks.
  Interventions: Biological: Lorigerlimab

INTERVENTIONS:
Biological: Lorigerlimab — Bispecific DART protein binding PD-1 and CTLA-4
  Other Names: MGD019

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, pharmacokinetics (PK) pharmacodynamics and preliminary antitumor activity of lorigerlimab.

This Phase 1, open-label study will characterize safety, dose-limiting toxicities (DLTs), and maximum tolerated/administered dose (MTD/MAD) of MGD019. Dose escalation will occur in a 3+3+3 design in patients with advanced solid tumors of any histology. Once the MTD/MAD is determined, a Cohort Expansion Phase will be enrolled to further characterize safety and initial anti-tumor activity in patients with specific tumor types anticipated to be sensitive to dual checkpoint blockade.

ELIGIBILITY:
Inclusion Criteria:

* Dose escalation: Patients with histologically proven, unresectable, locally advanced or metastatic solid tumors for whom no approved therapy with demonstrated clinical benefit is available or patients who are intolerant to standard therapy.
* Cohort Expansion Phase:
* Checkpoint inhibitor-naïve squamous cell NSCLC, including:

  1. Patients that have progressed during or following treatment with platinum-based chemotherapy for advanced disease. Patients harboring an activating epidermal growth factor receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) rearrangement must have progressed following at least one available EGFR or ALK targeted therapy. ROS1 rearrangement or BRAF mutation must have progressed following at least 1 available EGFR (including osimertinib for EGFR T790M-mutated NSCLC), ALK, ROS1 or BRAF targeted therapy, respectively
  2. Patients that have progressed during or following treatment with platinum-based chemotherapy for advanced disease and patients with previously untreated squamous cell NSCLC without activating mutations for whom checkpoint inhibitor therapy is not approved or available.
* Advanced non-microsatellite instability-high colorectal cancer (CRC) with recurrence, progression, or intolerance to standard therapy consisting of at least 2 prior standard regimens. CRC harboring an activating EGFR mutation must have progressed during or following at least one available EGFR targeted therapy. Patients who are inappropriate candidates for or have refused treatment with these regimens are also eligible. Patients should have received no more than 4 prior lines of systemic therapy.
* Checkpoint inhibitor-naïve mCRPC that has progressed during or following no more than 2 prior lines of an androgen receptor antagonist or androgen synthesis inhibitor (e.g., enzalutamide or abiraterone, respectively), if approved and available, with a PSA value of at least 2 ng/mL and meeting at least one of the following:
* Progression in measurable disease (RECIST v1.1).
* Appearance of 2 or more new bone lesions according to Prostate Cancer Working Group 2 (PCWG-2).
* Rising PSA defined as at least two sequential rises in PSA.
* Eligible patients may have received prior chemotherapy (i.e. docetaxel), and patients with known homologous recombination (HRR) pathway gene alterations must have received the applicable approved therapy (e.g. olaparib).
* Cutaneous melanoma that has progressed during or following systemic treatment for unresectable, locally advanced, or metastatic disease. Patients will have received PD-(L)1 and/or CTLA-4 pathway inhibitors where available and indicated.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy ≥ 12 weeks.
* Measurable disease as per RECIST 1.1 for the purpose of response assessment must either (a) not reside in a field that has been subjected to prior radiotherapy or (b) have demonstrated clear evidence of radiographic progression since the completion of prior radiotherapy and prior to study enrollment.
* All patients must have an identified formalin-fixed, paraffin embedded (FFPE) tumor specimen (up to 20 slides or a block) for immunohistochemical evaluation of pharmacodynamic markers of interest. Patients may undergo a fresh tumor biopsy during the screening period if a tumor sample is not available. Patients in the mCRPC expansion cohort with bone only disease not amenable to fresh biopsy may be eligible in consultation with the Sponsor.
* Acceptable laboratory parameters and adequate organ reserve.

Exclusion Criteria:

* In patients who have previously received an immune checkpoint inhibitor (e.g., anti-PD-L1, anti-PD-1, anti-CTLA-4), toxicities related to the checkpoint inhibitor must have resolved to ≤ Grade 1 or baseline. Patients with well controlled immune endocrinopathies secondary to prior checkpoint therapy are eligible.
* Patients with symptomatic CNS metastases. Patients with history of prior CNS metastasis must have been treated, must be asymptomatic, and must not have concurrent treatment for the CNS disease, progression of CNS metastases on magnetic resonance imaging (MRI) or computed tomography (CT) for at least 14 days after last day of prior therapy for the CNS metastases, or concurrent leptomeningeal disease or cord compression.
* Patients who sustained the following Grade 3 immune checkpoint inhibitor related AEs are ineligible: Ocular AE, changes in liver function tests that met the criteria for Hy's law (> 3 × ULN of either ALT or AST with concurrent > 2 × ULN of total bilirubin and without alternate etiology), neurologic toxicity, colitis, renal toxicity, pneumonitis.
* Patients who have received prior therapy with a combination of monoclonal antibodies against PD-1/PD-L1 and CTLA-4 will be excluded in the Cohort Expansion (this does not apply to the melanoma expansion cohort).
* Patients with any history of known or suspected autoimmune disease with certain exceptions
* History of prior allogeneic bone marrow, stem-cell, or solid organ transplantation.
* History of trauma or major surgical procedure within 4 weeks prior to initiation of study drug administration.
* Systemic antineoplastic therapy, or investigational therapy (for all tumor types) or androgen receptor antagonist/androgen synthesis inhibitor for mCRPC (e.g., enzalutamide or abiraterone, respectively) within the 4 weeks prior to initiation of study drug administration.
* Treatment with radiation therapy within 2 weeks prior to initiation of study drug administration.
* Radioligand (e.g., radium-223) within 6 months prior to initiation of study drug administration for mCRPC in the Cohort Expansion Phase.
* Serum testosterone > 50 ng/dl or > 1.7 nmol/L for mCRPC in the Cohort Expansion Phase.
* Confirmed or presumed COVID-19/SARS-CoV-2 infection. While SARS-CoV-2 testing is not mandatory for study entry, testing should follow local clinical practice guidelines/standards. Patients with a positive test result for SARS-CoV-2 infection, known asymptomatic infection, or presumed infection are excluded. Patients may be considered eligible after a resolved SARS-CoV-2 infection once he or she remains afebrile for at least 72 hours and after other SARS-CoV-2-related symptoms have fully recovered to baseline for a minimum of 72 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events | 30 days after last dose
  Safety is based on evaluation of adverse events (AEs) and serious adverse events (SAEs) from the time of study drug administration through the End of Study visit.

SECONDARY OUTCOMES:
Cmax | up to 108 weeks
  Maximum Plasma Concentration of lorigerlimab
Tmax | up to 108 weeks
  Time to reach maximum (peak) plasma concentration of lorigerlimab
AUC | up to 108 weeks
  Area Under the Plasma Concentration versus Time Curve of lorigerlimab
Ctrough | up to 108 weeks
  Trough plasma concentration of lorigerlimab
CL | up to 108 weeks
  Total body clearance of the drug from plasma of lorigerlimab
Vss | up to 108 weeks
  Apparent volume of distribution at steady state of lorigerlimab
t1/2 | up to 108 weeks
  Terminal half life of lorigerlimab
Percent of patients with anti-drug antibodies against lorigerlimab | up to 108 weeks
  Immunogenicity
Objective response rate (ORR) | Every 12 weeks, up to 4 years
  The number of participants who have a complete response (CR) or partial response (PR) to treatment. Efficacy assessed using conventional Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1)
Duration of Response (DoR) | Every 12 weeks until withdrawal of consent, lost to follow up, death, or end of the study, up to 4 years
  DoR is defined as the time from the date of initial response (CR or PR) to the date of first documented PD or death from any cause, whichever occurs first
Progression free survival (PFS) | Tumor status assessed every 12 weeks. Survival status is assessed approximately every 12 weeks after the last dose of study treatment until withdrawal of consent, lost to follow up, death, or end of the study, up to 4 years
  PFS is defined as the time from the first dose date to the date of first documented PD or death from any cause, whichever occurs first.
Overall survival (OS) | OS status is assessed approximately every 12 weeks after the last dose of study treatment until withdrawal of consent, lost to follow up, death, or end of the study, up to 4 years
  OS is defined as the time from the first dose date to the date of death from any cause.
Prostate specific antigen (PSA) response rate in mCRPC | Every 3 weeks on treatment, then every 3 months up to 2 years post last treatment
  Percent of patients with 50% or more decline in PSA and confirmed 3 weeks later
Best PSA percent change in mCRPC | Every 3 weeks on treatment, then every 3 months up to 2 years post last treatment
  Best percent change in PSA from baseline
Duration of PSA response | Every 3 weeks on treatment, then every 3 months up to 2 years post last treatment
  Time from PSA response to time of PSA progression
Radiographic progression-free survival (PFS) in metastatic castration-resistant prostate cancer (mCRPC) | up to 2 years post last treatment
  Time from first dose to first occurrence of radiographic progression, or death
Time to PSA progression in mCRPC | PSA is assessed every 3 weeks while on treatment, every 3 months for up to 2 years post-treatment
  The time from the first dose of MGD019 to the first documented PSA progression. PSA progression is defined as an increase that is ≥ 25% and ≥ 2 ng/mL the baseline or lowest value observed, and which confirmed by a second value at least 3 weeks later

CONTACTS AND LOCATIONS:
Overall Officials: Denise Casey, MD, Study Director — MacroGenics
Locations (39):
- United States (17):
  - University of Chicago Medical Center, Chicago, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Oncology Hematology West p.c. dba Nebraska Cancer Specialists, Grand Island, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Providence Portland Medical Center, Portland, Oregon
  - UPMC Hillman Cancer Center, Camp Hill, Pennsylvania
  - UPMC Hillman Cancer Center, Carlisle, Pennsylvania
  - UPMC Hillman Cancer Center, Erie, Pennsylvania
  - UPMC Pinnacle Harrisburg, Harrisburg, Pennsylvania
  - UPMC Pinnacle - Community Osteopathic Medical Sciences Pavilion (MSP), Harrisburg, Pennsylvania
  - UPMC Pinnacle - Ortenzio Cancer Center (OCC), Mechanicsburg, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - UPMC Hillman Cancer Center at UPMC Memorial, York, Pennsylvania
  - The Sarah Cannon Research Institute / Tennessee Oncology, Nashville, Tennessee
- Bulgaria (5):
  - Complex Oncology Center - Burgas" EOOD, Department of Medical Oncology, Burgas
  - Multiprofile Hospital for Active Treatment-Uni Hospital, Panagyurishte
  - Multiprofile Hospital for Active Treatment "Heart and Brain"" EAD, Clinic of Medical Oncology, Pleven
  - Complex Oncology Center - Ruse EOOD, Rousse
  - University Mulitprofile Hospital for Active Treatment "Sv. Ivan Rilski, Sofia
- Poland (7):
  - University Clinical Centre, Early Clinical Trials Unit, Gdansk
  - Pratia MCM Krakow, Krakow
  - Europejskie Centrum Zdrowia Otwock, Otwock
  - Med-Polonia Sp. z.o.o., Poznan
  - LUX MED Onkologia Sp. z.o.o., Warsaw
  - Narodowy Instytut Onkologii im, Warsaw
  - Mazovian Onkological Hospital, Wieliszew
- Spain (3):
  - ICO Badalona / Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario La Princesa, Madrid
- Ukraine (7):
  - Communal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro, Dnipro
  - Communal Non-Profit Enterprise "Regional Center of Oncology", Oncosurgical Department of Head and Neck, Kharkiv
  - Communal Nonprofit Enterprise "Regional Clinical Oncology Center of Kirovohrad Regional Council", Kirovohrad
  - Kyiv City Clinical Oncological Centre, Kyiv
  - National Cancer Institute of Ukraine, Kyiv
  - Sumy Clinical Oncological Hospital, Sumy
  - Communal Nonprofit Enterprise "Podilsky Regional Center of Oncology", Vinnytsia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berezhnoy A, Sumrow BJ, Stahl K, Shah K, Liu D, Li J, Hao SS, De Costa A, Kaul S, Bendell J, Cote GM, Luke JJ, Sanborn RE, Sharma MR, Chen F, Li H, Diedrich G, Bonvini E, Moore PA. Development and Preliminary Clinical Activity of PD-1-Guided CTLA-4 Blocking Bispecific DART Molecule. Cell Rep Med. 2020 Dec 22;1(9):100163. doi: 10.1016/j.xcrm.2020.100163. eCollection 2020 Dec 22. PMID 33377134
- See also: Link to published 2020 manuscript — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7762776/